CLINICAL TRIAL: NCT00467311
Title: Diagnostic, Transversal, Comparative, Not Randomized Trial for the Evaluation of Cystatin C as an Early Marker of Contrast-Medium Nephropathy in High-and-Intermedium-Risk Patients Undergoing to Cardiac Catheterization
Brief Title: Cystatin C as an Early Marker of Contrast-Medium Nephropathy in Cardiac Catheterization Patients
Status: Completed | Type: Observational
Sponsor: National Heart Institute, Mexico (Other Government)
Other Study IDs: 07552
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Contrast Induced Nephropathy; Acute Renal Failure
Keywords: Contrast-induced nephropathy; Cystatin C; Contrast media; Creatinine; Cardiac Catheterization
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis:

Cystatin C compared with creatinine is a better and earlier marker of contrast-induced nephropathy in high and intermedium risk cardiac catheterization patients.

Primary Objective:

Establish if Cystatin C is superior detecting contrast-induced nephropathy than creatinine in high and intermedium risk cardiac catheterization patients.

DETAILED DESCRIPTION:
Contrast induced-nephropathy is a complication that is underestimated in clinical practice after cardiac catheterization. During the last 30 years, because of the increasing use of contrast medium for diagnostic and therapeutic procedures, this has become the third in-hospital cause of acute renal failure (12%). That's why, it is necessary to establish an earlier marker of renal dysfunction that can help us in the diagnosis and allow us to initiate the appropriate therapeutics, because depending on the severity of the renal damage, it can increase the cardiovascular risk and morbidity.

The risk of contrast medium nephropathy is still present even with the use of low osmolarity contrast media, and many patients increase their in-hospital days, costs and hemodialysis requirement.

Cystatin C is a non glucosylated protein produced in nucleated cells in a constant rate, and because of its low molecular weight it's filtered through the glomerular membrane without restriction and it's fully reabsorbed in the proximal tubule, that's why it's considered an excellent marker evaluating the glomerular filtration rate in patients with acute renal failure during the first 24-48 hours.

We propose that Cystatin C can be useful as an earlier and superior marker of contrast-induced nephropathy in high and intermedium cardiac catheterization patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 20 years old
* Indication for coronariography and/or percutaneous coronary intervention
* Voluntary written consent for the realization of coronariography and/or percutaneous intervention and for the participation in this clinical trial
* A MEHRAN contrast-induced nephropathy score from six to fifteen.

Exclusion Criteria:

* N-Acetylcystein and Fenoldopam pre-medication
* Low risk patients according MEHRAN classification
* Cardiogenic and septic shock
* Acute renal failure by any other cause
* Patients with chronic kidney failure requiring any kind of dialysis
* Patients unable to complete follow-up
* Exposure to contrast media 48 hours prior to study
* Patients unable to give consent
* Receiving contrast media other than non-ionic

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 20 years old with an indication for coronariography and/or percutaneous coronary intervention, and with a MEHRAN contrast-induced nephropathy score from six to fifteen.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jhonathan L Uribe-González, MD, MSc, Principal Investigator — Ignacio Chávez National Institute of Cardiology; Jorge G Hernández, MD, FSCAI, Study Chair — Ignacio Chávez National Institute of Cardiology; Marco A Martínez-Rios, Study Director — Ignacio Chávez National Institute of Cardiology; Marco A Peña-Duque, MD, Principal Investigator — Ignacio Chávez National Institute of Cardiology
Locations (1):
- Ignacio Chávez National Institute of Cardiology, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Goldenberg I, Matetzky S. Nephropathy induced by contrast media: pathogenesis, risk factors and preventive strategies. CMAJ. 2005 May 24;172(11):1461-71. doi: 10.1503/cmaj.1040847. PMID 15911862
- [Background] Rickli H, Benou K, Ammann P, Fehr T, Brunner-La Rocca HP, Petridis H, Riesen W, Wuthrich RP. Time course of serial cystatin C levels in comparison with serum creatinine after application of radiocontrast media. Clin Nephrol. 2004 Feb;61(2):98-102. doi: 10.5414/cnp61098. PMID 14989628
- [Background] Schuck O, Teplan V, Jabor A, Stollova M, Skibova J. Glomerular filtration rate estimation in patients with advanced chronic renal insufficiency based on serum cystatin C levels. Nephron Clin Pract. 2003;93(4):c146-51. doi: 10.1159/000070234. PMID 12759583
- [Background] Han WK, Bonventre JV. Biologic markers for the early detection of acute kidney injury. Curr Opin Crit Care. 2004 Dec;10(6):476-82. doi: 10.1097/01.ccx.0000145095.90327.f2. PMID 15616389
- [Background] Villa P, Jimenez M, Soriano MC, Manzanares J, Casasnovas P. Serum cystatin C concentration as a marker of acute renal dysfunction in critically ill patients. Crit Care. 2005 Apr;9(2):R139-43. doi: 10.1186/cc3044. Epub 2005 Feb 7. PMID 15774046
- [Background] Shlipak MG, Sarnak MJ, Katz R, Fried LF, Seliger SL, Newman AB, Siscovick DS, Stehman-Breen C. Cystatin C and the risk of death and cardiovascular events among elderly persons. N Engl J Med. 2005 May 19;352(20):2049-60. doi: 10.1056/NEJMoa043161. PMID 15901858
- [Background] Lameire N, Hoste E. Reflections on the definition, classification, and diagnostic evaluation of acute renal failure. Curr Opin Crit Care. 2004 Dec;10(6):468-75. doi: 10.1097/01.ccx.0000144939.24897.71. No abstract available. PMID 15616388
- [Background] Loew M, Hoffmann MM, Koenig W, Brenner H, Rothenbacher D. Genotype and plasma concentration of cystatin C in patients with coronary heart disease and risk for secondary cardiovascular events. Arterioscler Thromb Vasc Biol. 2005 Jul;25(7):1470-4. doi: 10.1161/01.ATV.0000168416.74206.62. Epub 2005 Apr 28. PMID 15860739
- [Background] Mares J, Stejskal D, Vavrouskova J, Urbanek K, Herzig R, Hlustik P. Use of cystatin C determination in clinical diagnostics. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2003 Dec;147(2):177-80. PMID 15037900
- [Background] Hoek FJ, Kemperman FA, Krediet RT. A comparison between cystatin C, plasma creatinine and the Cockcroft and Gault formula for the estimation of glomerular filtration rate. Nephrol Dial Transplant. 2003 Oct;18(10):2024-31. doi: 10.1093/ndt/gfg349. PMID 13679476
- [Background] Bokenkamp A, Domanetzki M, Zinck R, Schumann G, Byrd D, Brodehl J. Cystatin C--a new marker of glomerular filtration rate in children independent of age and height. Pediatrics. 1998 May;101(5):875-81. doi: 10.1542/peds.101.5.875. PMID 9565418
- [Background] Herget-Rosenthal S, Marggraf G, Husing J, Goring F, Pietruck F, Janssen O, Philipp T, Kribben A. Early detection of acute renal failure by serum cystatin C. Kidney Int. 2004 Sep;66(3):1115-22. doi: 10.1111/j.1523-1755.2004.00861.x. PMID 15327406
- [Background] Coll E, Botey A, Alvarez L, Poch E, Quinto L, Saurina A, Vera M, Piera C, Darnell A. Serum cystatin C as a new marker for noninvasive estimation of glomerular filtration rate and as a marker for early renal impairment. Am J Kidney Dis. 2000 Jul;36(1):29-34. doi: 10.1053/ajkd.2000.8237. PMID 10873868
- [Background] O'Riordan SE, Webb MC, Stowe HJ, Simpson DE, Kandarpa M, Coakley AJ, Newman DJ, Saunders JA, Lamb EJ. Cystatin C improves the detection of mild renal dysfunction in older patients. Ann Clin Biochem. 2003 Nov;40(Pt 6):648-55. doi: 10.1258/000456303770367243. PMID 14629803
- See also: National Institute of Cardiology — http://www.cardiologia.org.mx